CLINICAL TRIAL: NCT05442853
Title: Continuous Glucose Monitoring for Hyperglycemia in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malcom Randall VA Medical Center (U.S. Federal Agency)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Andrew Franck, Primary Investigator, Malcom Randall VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202201063
Record Dates: First submitted 2022-06-16; First posted 2022-07-05 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Hyperglycemia; Hypoglycemia; Critical Illness; Diabetes Mellitus
MeSH Terms: conditions — Hyperglycemia; Hypoglycemia; Critical Illness; Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Continuous Glucose Monitoring (Active Comparator): Study subjects in this arm will receive glycemic management based on continuous glucose monitoring with CGM device. CGM readings will be available to patients, nurses, and the treating team. All treatment decisions for this group will be based on CGM readings, confirmatory POC readings (as necessary), and venipuncture.
  Interventions: Device: Continuous glucose monitoring
- Point of Care Glucose Monitoring (Active Comparator): Study subjects in this arm will receive glycemic management based on point of care blood glucose readings. CGM will be placed in blinded mode and used for study comparison only. Patients, nurses, and other treatment team will be blinded to the CGM readings. All treatment decisions for this group will be based on POC readings and venipuncture
  Interventions: Device: Point of care glucose monitoring

INTERVENTIONS:
Device: Continuous glucose monitoring — Continuous glucose monitoring involves a wearable device that measures glucose with a sensor that is inserted subcutaneously. The sensor transmits data to receiving device that displays the glucose values.
  Arms: Continuous Glucose Monitoring
Device: Point of care glucose monitoring — Point of care glucose monitoring involves use of an external device that can provide glucose readings at a patient's bedside. These devices require a small blood sample from venous, arterial, or capillary fingerstick blood. The blood sample is analyzed by the device and reports a glucose value within 5 minutes. This method of glucose monitoring is a mainstay and standard of care for most hospitals in the United States.
  Arms: Point of Care Glucose Monitoring

SUMMARY:
The investigators intend to conduct a single-center, prospective, randomized comparative trial of patients admitted to the intensive care unit (ICU) who received continuous glucose monitoring (CGM) vs point of care (POC) glucose monitoring. The study will examine relevant outcomes for patients in the ICU with diabetes mellitus and/or hyperglycemia. The primary outcome of the study will be the proportion of time in target range (blood glucose 70-180 mg/dL).

DETAILED DESCRIPTION:
Study Purpose:

The purpose of this study is to compare the use of continuous glucose monitoring (CGM) versus point of care (POC) glucose monitoring in the intensive care unit (ICU) setting for differences in glycemic control and other important outcomes.

Research Plan:

This will be a prospective, single-center, randomized comparative trial of adult patients at North Florida/South Georgia Veterans Health System anticipated to be admitted to an ICU for a minimum of 48 hours after enrollment. Study participants will be randomly assigned to one of the study groups (CGM or POC) after being found eligible for inclusion and giving consent to participate. The CGM group will receive glycemic management based on CGM readings. The POC group will receive glycemic management based on POC glucose readings.

Study Outcomes:

Groups will be compared for differences in clinical and safety outcomes. The primary outcome will be the proportion of time in target range (BG 70-180mg/dL). Secondary outcomes will include mean glucose, hypoglycemia, hyperglycemia, ICU length of stay, mortality, glucose variability, cost, and patient satisfaction. Safety outcomes will include new infection, acute kidney injury, delirium, agitation, and pain.

Analysis Methods:

Descriptive statistics and inferential statistical methods will be used as appropriate to report findings of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-89
* Past medical history of any diabetes mellitus OR patients with at least 1 measured BG of 180 being treated with insulin (subcutaneous or infusion)
* Enrollment will occur within 72 hours after being admitted to an ICU if history of diabetes
* Enrollment will occur within 72 hours after developing hyperglycemia in ICU if no diabetes

Exclusion Criteria:

* Pregnant patients
* Patients using CGMs in the outpatient setting
* Diagnosis of diabetic ketoacidosis (DKA)
* Diagnosis of hyperosmolar hyperglycemic state (HHS)
* Anticipated to require prone positioning while on insulin therapy
* Any contraindications to CGMs based on manufacturer labeling
* BG above maximum reading for CGM (e.g. greater than 400 mg/dL)
* Receiving medication that could interfere with CGM readings (based on manufacturer specifications)
* Receiving any dose of hydroxyurea as this could falsely elevate the sensor readings (if applicable for specific CGM)
* Receiving greater than 1,000mg acetaminophen every 6 hours in any form as this could falsely elevate the sensor readings (if applicable for specific CGM)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Franck, PharmD, Principal Investigator — US Department of Veterans Affairs
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franck AJ, Hendrickson AL, Telford ED, Davids BL, Murray Casanova I, Rosen AN, Hadigal S, Ross RC. Continuous Glucose Monitoring for Hyperglycemia in Critically Ill Patients: A Randomized Controlled Trial. Chest. 2025 Aug;168(2):326-335. doi: 10.1016/j.chest.2025.02.006. Epub 2025 Feb 15. PMID 39956190

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Started | 43 | 42
Completed | 43 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 75 [69 to 76.5] | 72 [67.3 to 76.8] | 74 [67.5 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 43 | 42 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 42 | 42 | 84
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 38 | 32 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Time in Target Blood Glucose Range (BG 70-180mg/dL)
Description: Percentage of time within time glucose range based on CGM readings
Time Frame: For duration of study enrollment (up to 10 days)
Measure: Mean (Standard Deviation); unit: percentage of time within target range
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
percentage of time within target range | 60.5 (30.5) | 61.4 (28.3)

2. Secondary Outcome: Time in Clinically Significant Hypoglycemic Range (BG < 54 mg/dL)
Description: Percentage of time with BG less than 54 mg/dl as measured by CGM
Time Frame: For duration of study enrollment (up to 10 days)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
percentage of time | 0.2 (1.0) | 1.1 (3.1)

3. Secondary Outcome: Time in Hypoglycemic Range (BG 54-69 mg/dL)
Description: Percentage of time in this glucose range as measured by CGM
Time Frame: For duration of study enrollment (up to 10 days)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
percentage of time | 1.4 (6.8) | 0.9 (2.0)

4. Secondary Outcome: Time in Hyperglycemic Range (BG 181-250 mg/dL)
Description: Percentage of time in this glucose range as measured by CGM
Time Frame: For duration of study enrollment (up to 10 days)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
percentage of time | 29.6 (24.4) | 25.6 (17.0)

5. Secondary Outcome: Time in Clinically Relevant Hyperglycemic Range (BG >250 mg/dL)
Description: Percentage of time in this glucose range as measured by CGM
Time Frame: For duration of study enrollment (up to 10 days)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
percentage of time | 8.0 (14.6) | 11.0 (18.4)

6. Secondary Outcome: ICU Length of Stay
Description: Total time (in days or hours) in the intensive care unit
Time Frame: At time of ICU discharge or death (assessed up to 1 month)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
days | 3.9 (2.8) | 4.6 (3.8)

7. Secondary Outcome: ICU Mortality
Description: Death from any cause during ICU stay
Time Frame: At time of ICU discharge or death (assessed up to 1 month)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
Participants | 3 | 2

8. Secondary Outcome: 30 Day Mortality
Description: Death from any cause at 30 days after admission to the ICU
Time Frame: At 30 days or time of death
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
Participants | 8 | 2

9. Secondary Outcome: Cost Associated With Monitoring
Description: Monetary value assigned to blood glucose monitoring
Time Frame: For duration of study enrollment (up to 10 days)
Measure: Number; unit: dollars
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
dollars | 0 | 0

10. Secondary Outcome: Mean Blood Glucose
Description: Average blood glucose (< 180 mg/dl) during the study timeframe
Time Frame: For duration of study enrollment (up to 10 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
Participants | 28 | 27

11. Secondary Outcome: Glucose Variability
Description: a. % coefficient of variation = SD/mean BG*100%
Time Frame: For duration of study enrollment (up to 10 days)
Measure: Mean (Standard Deviation); unit: percentage of variability
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
percentage of variability | 21.0 (6.9) | 22.3 (7.2)

12. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction with glucose monitoring as assessed by survey on Likert Scale (1-5). Score of 1 being 'very dissatisfied' to score of 5 being 'very satisfied.'
Time Frame: Once at completion of study enrollment (at day 10 or sooner)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
score on a scale | 5 [4 to 5] | 4 [3 to 4]

13. Secondary Outcome: New Infection
Description: Any infection diagnosis that was not present upon admission to the ICU
Time Frame: Assessed daily, For duration of study enrollment (up to 10 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
Participants | 2 | 2

14. Secondary Outcome: New Acute Kidney Injury
Description: New acute kidney injury (based on Acute Kidney Injury Network guideline definitions) not present upon admission to the ICU
Time Frame: Assessed daily, For duration of study enrollment (up to 10 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
Participants | 6 | 4

15. Secondary Outcome: ICU Delirium
Description: Development of ICU delirium, based on Confusion Assessment Method for the ICU (CAM-ICU) score, with any positive score indicating presence of delirium.
Time Frame: Assessed daily, For duration of study enrollment (up to 10 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
Participants | 1 | 1

16. Secondary Outcome: Agitation
Description: Richmond agitation scores (-5 to +4), with scores of +2 or more indicated agitation.
Time Frame: Assessed daily, For duration of study enrollment (up to 10 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
Participants | 2 | 1

17. Secondary Outcome: Pain Associated With Glucose Monitoring
Description: Patient reported pain associated with glucose monitoring
Time Frame: Assessed daily, For duration of study enrollment (up to 10 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
Number analyzed (Participants) | 43 | 42
Participants | 1 | 4

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: up to 30 days after admission to the ICU. Serious and Other Adverse Events: for duration of study enrollment (up to 10 days)
Arm/Group | Continuous Glucose Monitoring | Point of Care Glucose Monitoring
All-Cause Mortality (participants affected / at risk) | 8/43 | 2/42
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 2/43 | 1/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Glucose Monitoring (N=43) | Point of Care Glucose Monitoring (N=42)
Inability to accurately calibrate CGM (Product Issues) | 2 (2) | 0 (0)
Minor Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT05442853/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT05442853/ICF_001.pdf